CLINICAL TRIAL: NCT02236949
Title: Sustainability of a Multidimensional Knowledge Translation Intervention to Improve Paediatric Pain Practices and Outcomes
Brief Title: Sustainability of a Knowledge Translation Intervention to Improve Paediatric Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Bonnie Stevens, Bonnie Stevens RN PhD, Signy Hildur Eaton Chair in Paediatric Nursing, Associate Chief of Nursing Research, Senior Scientist Research Institute, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1000026324
Record Dates: First submitted 2014-09-05; First posted 2014-09-11 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Pain
Keywords: pediatric pain; intervention sustainability
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pain Practice Change Booster (Experimental): Pain Practice Change Booster Intervention: 12 months after the EPIQ intervention, and every 4 months for 2 years, a 30-60 minute standardized booster session was delivered to a small group of champions in each hospital unit randomized to the intervention group. Two co-facilitators familiar with the EPIQ intervention conducted all booster sessions via teleconference. Booster sessions included reviewing the effectiveness knowledge translation strategies champions implemented over the past four months to sustain and improve targeted pain practices; determining the sustainability of the pain practice changes, developing a commitment to change plan of action for the next four months.
  Interventions: Behavioral: Pain Practice Change Booster Intervention
- Usual Care Group (No Intervention): No interventions associated with the study were conducted on these units.

INTERVENTIONS:
Behavioral: Pain Practice Change Booster Intervention — See experimental arm for a description of the intervention
  Arms: Pain Practice Change Booster

SUMMARY:
The purpose of this research study is to evaluate the effectiveness of short refresher sessions. "Pain Practice Change Boosters" given at regular intervals to sustain improved pain process (assessment and management) and clinical outcomes (pain intensity) achieved during a 15 month knowledge translation intervention, Evidence-based Practice for Improving Quality (EPIQ), in 8 children's hospitals in Canada; and to determine the factors that affect that sustainability. The CIHR Team in Children's Pain (2006-2011) evaluated the effectiveness of the EPIQ intervention in 32 hospital units (4 units at each hospital site). 16 hospital units were allocated to the intervention group and 16 units continued with standard care. The current study focuses on the 16 hospital units that implemented the EPIQ intervention only.

DETAILED DESCRIPTION:
This is an 8 hospital repeated measures Randomized Controlled Trial design using a centrally controlled cluster random allocation of units with stratification by hospital. The sample consisted of the 16 hospital units that implemented the EPIQ intervention in the CIHR Team in Children's Pain study. Randomization was restricted so there was one intervention unit and one standard care unit at each site. Outcomes were measured at 3 time points:12 months after the completion of the EPIQ intervention: Baseline (Time 1); 12 months following the implementation of the Booster intervention (Time 2); and 36 months following the implementation of the Booster intervention (Time 3), including the frequency and proportion of children receiving pain assessment and management strategies, children's pain intensity during painful procedures, and health care professionals' perceptions of the context of sustainability.

ELIGIBILITY:
Inclusion Criteria:

Hospitals met the following inclusion criteria in at least four patient care units:

* distinct geographic location and administrative structure;
* minimum of 15 beds per unit;
* care for children exposed to painful procedures for diagnostic or therapeutic purposes; and
* implementation of pharmacological and non-pharmacological interventions to manage pain.

The 16 participating hospital units had implemented the EPIQ intervention in the CIHR Team in Children's Pain study. Patients in the participating hospital units were eligible to be included in the determination of the pain practice and clinical outcomes if they:

* were between 32 weeks gestational age at birth and 18 years;
* received skin breaking procedures; and
* were admitted to the unit for >24 hours.

Surveys used to determine factors influencing sustainability were administered to health care professionals in all participating units, who had at least 1 year of professional experience, had worked on the unit for at least 6 months, and spoke English or French.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3907 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pain Process Outcomes (pain assessment) | T1 (Baseline)
  Pain process outcomes included the proportion of children per unit whose pain was assessed and whether a validated pain measure was used. Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).
Factors Influencing Sustainability: The Alberta Context Tool (ACT) | T1 (Baseline)
  The Alberta Context Tool (ACT) (Estabrooks, 2011) was used to determine the factors that influence sustainability in each of the 16 participating hospital units, including organizational culture, leadership, readiness to change, organizational complexity, professional autonomy and support within the workplace. The ACT measures health care professionals' perceptions of these contextual factors at the unit and institutional levels. The tool was administered in survey form to staff on the participating units at 3 time points.
Pain Process Outcomes (pain assessment) | T2 (12 months following the implementation of the Booster)
  Pain process outcomes included the proportion of children per unit whose pain was assessed and whether a validated pain measure was used. Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).
Pain Process Outcomes (pain assessment) | T3 (24 months following the implementation of the Booster)
  Pain process outcomes included the proportion of children per unit whose pain was assessed and whether a validated pain measure was used. Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).
Factors Influencing Sustainability: The Alberta Context Tool (ACT) | T2 (12 months following the implementation of the Booster)
  The Alberta Context Tool (ACT) was used to determine the factors that influence sustainability in each of the 16 participating hospital units, including organizational culture, leadership, readiness to change, organizational complexity, professional autonomy and support within the workplace. The ACT measures health care professionals' perceptions of these contextual factors at the unit and institutional levels. The tool was administered in survey form to staff on the participating units at 3 time points.
Factors Influencing Sustainability: The Alberta Context Tool (ACT) | T3 (24 months following the implementation of the Booster)
  The Alberta Context Tool (ACT) was used to determine the factors that influence sustainability in each of the 16 participating hospital units, including organizational culture, leadership, readiness to change, organizational complexity, professional autonomy and support within the workplace. The ACT measures health care professionals' perceptions of these contextual factors at the unit and institutional levels. The tool was administered in survey form to staff on the participating units at 3 time points.
Pain Process Outcomes (pain management) | T1 (Baseline)
  Pain process outcomes included the proportion of children per unit who had painful procedures: (i) without pain management interventions, (ii) with pharmacological interventions, and (iii) with non-pharmacological interventions (i.e., physical or psychological). Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).
Pain Process Outcomes (pain management) | T2 (12 months following the implementation of the Booster)
  Pain process outcomes included the proportion of children per unit who had painful procedures: (i) without pain management interventions, (ii) with pharmacological interventions, and (iii) with non-pharmacological interventions (i.e., physical or psychological). Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).
Pain Process Outcomes (pain management) | T3 (24 months following the implementation of the Booster)
  Pain process outcomes included the proportion of children per unit who had painful procedures: (i) without pain management interventions, (ii) with pharmacological interventions, and (iii) with non-pharmacological interventions (i.e., physical or psychological). Data were collected from 30 patient charts on each unit for the previous 24 hours at 3 time points, using the Canadian Pediatric Pain Research (CPPR) database, which was used and validated in previous studies (Stevens, 2011, 2012, 2014).

SECONDARY OUTCOMES:
Clinical Pain Outcome: Pain Intensity | T1 (Baseline)
  Pain intensity was measured through patient observation during routinely scheduled painful procedures at 3 time points, using one of four validated, age-appropriate measures: Premature Infant Pain Profile (PIPP) (Stevens et al., 1996) Faces-Legs-Arms-Cry-Consolability Scale (FLACC) (Merkel et al., 1997), Faces Pain Scale-Revised (FPS-R) (Hicks et al., 2001), and Numerical Rating Scale (NRS) (Jensen et a., 1986). Data were collected by local pain experts, experienced pediatric clinicians, who were trained on the four measures to ensure accurate and standardized use.
Clinical Pain Outcome: Pain Intensity | T2 (12 months following the implementation of the Booster)
  Pain intensity was measured through patient observation during routinely scheduled painful procedures at 3 time points, using one of four validated, age-appropriate measures: Premature Infant Pain Profile (PIPP) (Stevens et al., 1996) Faces-Legs-Arms-Cry-Consolability Scale (FLACC) (Merkel et al., 1997), Faces Pain Scale-Revised (FPS-R) (Hicks et al., 2001), and Numerical Rating Scale (NRS) (Jensen et a., 1986). Data were collected by local pain experts, experienced pediatric clinicians, who were trained on the four measures to ensure accurate and standardized use.
Clinical Pain Outcome: Pain Intensity | T3 (24 months following the implementation of the Booster)
  Pain intensity was measured through patient observation during routinely scheduled painful procedures at 3 time points, using one of four validated, age-appropriate measures: Premature Infant Pain Profile (PIPP) (Stevens et al., 1996) Faces-Legs-Arms-Cry-Consolability Scale (FLACC) (Merkel et al., 1997), Faces Pain Scale-Revised (FPS-R) (Hicks et al., 2001), and Numerical Rating Scale (NRS) (Jensen et a., 1986). Data were collected by local pain experts, experienced pediatric clinicians, who were trained on the four measures to ensure accurate and standardized use.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Stevens, RN, PhD, Principal Investigator — The Hospital for Sick Children
Locations (7):
- Canada (7):
  - Stollery Chidlren's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Children's Hospital Winnipeg, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
  - CHU St. Justine, Montreal, Quebec

REFERENCES:
- [Background] Stevens BJ, Yamada J, Estabrooks CA, Stinson J, Campbell F, Scott SD, Cummings G; CIHR Team in Children's Pain. Pain in hospitalized children: Effect of a multidimensional knowledge translation strategy on pain process and clinical outcomes. Pain. 2014 Jan;155(1):60-68. doi: 10.1016/j.pain.2013.09.007. Epub 2013 Sep 8. PMID 24021861
- [Background] Stevens BJ, Harrison D, Rashotte J, Yamada J, Abbott LK, Coburn G, Stinson J, Le May S; CIHR Team in Children's Pain. Pain assessment and intensity in hospitalized children in Canada. J Pain. 2012 Sep;13(9):857-65. doi: 10.1016/j.jpain.2012.05.010. PMID 22958873
- [Background] Stevens BJ, Abbott LK, Yamada J, Harrison D, Stinson J, Taddio A, Barwick M, Latimer M, Scott SD, Rashotte J, Campbell F, Finley GA; CIHR Team in Children's Pain. Epidemiology and management of painful procedures in children in Canadian hospitals. CMAJ. 2011 Apr 19;183(7):E403-10. doi: 10.1503/cmaj.101341. Epub 2011 Apr 4. PMID 21464171
- [Background] Estabrooks CA, Squires JE, Hutchinson AM, Scott S, Cummings GG, Kang SH, Midodzi WK, Stevens B. Assessment of variation in the Alberta Context Tool: the contribution of unit level contextual factors and specialty in Canadian pediatric acute care settings. BMC Health Serv Res. 2011 Oct 4;11:251. doi: 10.1186/1472-6963-11-251. PMID 21970404
- [Derived] Stevens BJ, Yamada J, Promislow S, Barwick M, Pinard M; CIHR Team in Children's Pain. Pain Assessment and Management After a Knowledge Translation Booster Intervention. Pediatrics. 2016 Oct;138(4):e20153468. doi: 10.1542/peds.2015-3468. Epub 2016 Sep 1. PMID 27587614